CLINICAL TRIAL: NCT06358066
Title: Clinical Evaluation of Biomimetic Self -Assembling Peptide (p11-4) in The Remineralization of Early Enamel Caries in Permanent Teeth
Brief Title: The Remineralization of Early Enamel Caries in Permanent Teeth
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sara Ahmed Fathy Mohamed, principal investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: self assembling peptides
Record Dates: First submitted 2024-03-29; First posted 2024-04-10 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: White Spot Lesion
Keywords: Remineralization
MeSH Terms: interventions — Fluorides; Paint

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- curodont repair fluoride plus (Experimental): Group I (study group): Teeth will be treated with self-assembling peptide (P11-4) fluoride plus varnish.
  Interventions: Drug: self assembling peptide p11-4 with fluoride
- fluoride varnish (Active Comparator): Group II (control group): Teeth will be treated with fluoride varnish.
  Interventions: Drug: 5% sodium fluoride varnish

INTERVENTIONS:
Drug: self assembling peptide p11-4 with fluoride — Self-assembling peptide (P11-4) fluoride plus will be applied according to the manufacturer's instructions by pushing the two cylinders together and will left for 5 min till the tooth surface appears dry to insure its diffusion
  The remineralizing process of the early enamel carious lesions will be assessed quantitatively using the laser fluorescence DIAGNOdent measuring and assessed qualitatively using ICDAS II scoring system at baseline 1, 3, 6 months post-treatment
  Other Names: curodont repair fluoride plus varnish
  Arms: curodont repair fluoride plus
Drug: 5% sodium fluoride varnish — Fluoride varnish will be applied under manufacturer instructions by applying thin layer of varnish with a brush in strokes The remineralizing process of the early enamel carious lesions will be assessed quantitatively using the laser fluorescence DIAGNOdent measuring and assessed qualitatively using ICDAS II scoring system at baseline 1, 3, 6 months post-treatment
  Other Names: charm fluoride varnish
  Arms: fluoride varnish

SUMMARY:
Evaluate clinically the remineralizing potential of self-assembling peptide ( P11-4) fluoride plus in early enamel carious lesions of permanent anterior teeth.

DETAILED DESCRIPTION:
Study design This study will be conducted as a randomized controlled clinical trial. Study setting The study will be carried out in the clinic of Pediatric Dentistry Department, Faculty of Dentistry, Tanta University.

Group assignment:

Fifty children will be randomly allocated using simple random table into two groups as follows:

* Group I (study group): Teeth will be treated with self-assembling peptide (P11-4) fluoride plus varnish.
* Group II (control group): Teeth will be treated with fluoride varnish.

Ethical consideration The purpose of the present study will be explained to both the parents and children and informed consents will be obtained as well as ascents from children .The researcher will be obligated to do dental treatment for every child according to his-her condition as compensation according to the guidelines on human research adopted by the Research Ethics Committee, Faculty of Dentistry, Tanta University.

Materials to be used in the study:

Materials Composition Manufacture Trade names

Fluoride varnish

5% sodium fluoride (22.600ppm) Dentkist-korea Charm varnish R

Self-assembling peptide p11-4 Sodium Fluoride 0.05% Water,Chlorhexidine digluconate,Tromethamine, Trehalose Dihydrate, Oligopeptide-104, HydroxyPropyl MethylCellulose,Citric Acid,Sodium Hydroxide Credentis AG, Windisch, Switzerland CURODONT Repair ™ fluoride plus Polishing paste fluoride free Titanium Oxide Crosstex- Chicago,US Sparkle Free Prophy Paste

Methods

1. Clinical examination and assessments:

   * Full dental and medical history for the children will be recorded in the child chart.
   * Children will be examined under reflector light conditions using sterile mirrors and blunt end probes with compressed air.
   * Labial surface of one anterior tooth in each child will be cleaned and plaque debris will be removed using a prophylaxis paste fluoride free and a polishing brush 20,21,.
   * Early enamel carious Lesions will be assessed according to the International Caries Detection and Assessment System (ICDAS II; ranging between 1-3) and Laser fluorescence (LF) measurements DIAGNOdent* will be conducted and values will be recorded as baseline data22,23.
2. Clinical procedure:

   * The selected teeth will be isolated with rubber dam.
   * The labile surface of the teeth will be gently cleaned and dried with air syringe.
   * In Group I: Self-assembling peptide (P11-4) fluoride plus will be applied according to the manufacturer's instructions by pushing the two cylinders together and will left for 5 min till the tooth surface appears dry to insure its diffusion 15.
   * In Group II: Fluoride varnish will be applied under manufacturer instructions by applying thin layer of varnish with a brush in strokes 24.

   In all groups children will be advised to:
   * Not to rinse his or her mouth, eat, or drink for at least 30 minutes after the treatment, only soft food and drink can be consumed in the day of treatment 22.
   * The children use a soft toothbrush and fluoridated toothpaste as an oral hygiene regimen23.
3. Evaluation:

The remineralizing process of the early enamel carious lesions will be assessed qualitatively using ICDAS II scoring system (table 1) and quantitatively using the laser fluorescence DIAGNOdent measuring at baseline 1, 3, 6 months post-treatment

ELIGIBILITY:
Inclusion Criteria:

* Presence of active non-cavitated carious white spot lesions with DIAGNO/dent reading from 5 to 17 ,on labial surfaces of permanent anterior teeth and International Caries Detection And Assessment System II (ICDAS II) ranging between 1 and 3.
* The children' age range between 10 to14 years old.
* Children had completed fixed orthodontic treatment within the past week.
* Good oral hygiene with a plaque index score 0 or 1.
* No systemic diseases or medication affecting salivary flow.

Exclusion Criteria:

* Children with tetracycline pigmentation, dental fluorosis, or enamel hypoplasia.
* Children had fluoride application less than 3 months before the study.
* Presence of restoration and cavitation on the surface to be treated.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-06-06 (Estimated); Primary Completion 2024-11-06 (Estimated); Study Completion 2025-01-06 (Estimated)

PRIMARY OUTCOMES:
Remineralization potential | 1 month
  T0:baseline assessment --> T1:1 month(Application of Curodont repair flouride plus /fluoride varnish andAssessment of white spot lesion regression)--> T2: 3 months Assessment of white spot lesion regression__>T3: 6 months assessment of white spot lesion regression by: Inspection under magnification ICDAS II Score 0:Sound tooth surface:
  1. First visual change in enamel.
  2. Distinct visual change in enamel visible when wet, lesion must be visible when dry.
  by:Diagnodent

SECONDARY OUTCOMES:
Remineralization potential | 3 months
  [ Time Frame: T0:baseline assessment -->T1:1 month (Assessment of white spot lesion regression)--> T2:3 months(Application of Curodont repair flouride plus /fluoride varnish and Assessment of white spot lesion regression)--> T3: 6 months( Assessment of white spot lesion regression by Diagnodent , ICDASII

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of Dentistry,Tanta university, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 6 months